CLINICAL TRIAL: NCT03022994
Title: Duodenal and Rectal Histology in Non-celiac Wheat Sensitivity and Irritable Bowel Syndrome Patients
Status: Completed | Type: Observational
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Pasquale Mansueto, MD, University of Palermo
Other Study IDs: ACPM18
Record Dates: First submitted 2016-12-30; First posted 2017-01-18 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Non-celiac Wheat Sensitivity
Keywords: Non-celiac wheat sensitivity; eosinophils; lymphocytes; duodenal biopsies; rectal biopsies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biopsy specimens obtained from the bulb and the second duodenal portion and the rectum.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- NCWS patients: Forty consecutive adult patients with an IBS-like clinical presentation, according to Rome III criteria, and a definitive diagnosis of NCWS. The patients will be recruited between January 2016 and February 2017 at 2 centers: the Department of Internal Medicine at the University Hospital of Palermo, Italy, and the Department of Internal Medicine of the Hospital of Sciacca, Agrigento, Italy. All subjects will undergo upper gastrointestinal endoscopy and proctoscopy at the Gastroenterology Unit at the University Hospital of Palermo, Italy. Duodenal and rectal biopsies will be evaluated at 2 centers: the Pathology Unit at the University Hospital of Palermo, Italy, and the Institute of Pathology at the "Spedali Civili" of Brescia, Italy.
  Interventions: Other: Duodenum and rectum examination
- IBS patients: Forty sex- and age-matched subjects with IBS unrelated to NCWS or other food 'intolerance', diagnosed according to standard criteria during the same study period and enrolled, at the same 2 centers, as control group. All subjects will undergo upper gastrointestinal endoscopy and proctoscopy at the Gastroenterology Unit at the University Hospital of Palermo, Italy. Duodenal and rectal biopsies will be evaluated at 2 centers: the Pathology Unit at the University Hospital of Palermo, Italy, and the Institute of Pathology at the "Spedali Civili" of Brescia, Italy.
  Interventions: Other: Duodenum and rectum examination

INTERVENTIONS:
Other: Duodenum and rectum examination — All subjects will undergo upper gastrointestinal endoscopy and proctoscopy. In addition, it will be also evaluated duodenal and rectal biopsies.

SUMMARY:
Recently it has been reported that a consistent percentage of the general population consider themselves to be suffering from problems caused by wheat and/or gluten ingestion, even though they do not have CD or wheat allergy. This clinical condition has been named Non-Celiac Gluten Sensitivity' (NCGS). In a previous paper the investigators suggested the term 'Non-Celiac Wheat Sensitivity' (NCWS), since it is not known what component of wheat causes the symptoms in NCGS patients, and the investigators also showed that these patients had a high frequency of coexistent multiple food hypersensitivity. Nowadays only few data are available on the histological characteristic of duodenal and rectal biopsies of NCWS patients. The researchers have just demonstrated a significant eosinophils infiltration of the duodenal and colon mucosa, and a significant infiltration of CD45+/CD3-CD14- cells in the rectal mucosa of NCWS patients upon wheat challenge, thus configuring a diffuse gastrointestinal "inflammatory/immunologic" pattern. The aims of the present study are: 1) to investigate the histological characteristics in duodenal and rectal biopsies between NCWS and irritable bowel syndrome (IBS) patients, and 2) to evaluate which site (i.e. duodenal or rectal) shows "inflammatory/allergic" features useful for NCWS histological diagnosis.

DETAILED DESCRIPTION:
Recently it has been reported that a consistent percentage of the general population consider themselves to be suffering from problems caused by wheat and/or gluten ingestion, even though they do not have CD or wheat allergy. This clinical condition has been named Non-Celiac Gluten Sensitivity' (NCGS). In a previous paper the investigators suggested the term 'Non-Celiac Wheat Sensitivity' (NCWS), since it is not known what component of wheat causes the symptoms in NCGS patients, and the investigators also showed that these patients had a high frequency of coexistent multiple food hypersensitivity. The clinical picture of NCWS is characterized by combined gastrointestinal (bloating, abdominal pain, diarrhea and/or constipation, nausea, epigastric pain, gastroesophageal reflux, aphthous stomatitis) and extra-intestinal and/or systemic manifestations (headache, depression, anxiety, 'foggy mind,' tiredness, dermatitis or skin rash, fibromyalgia-like joint/muscle pain, leg or arm numbness, and anemia). Nowadays only few data are available on the histological characteristic of duodenal and rectal biopsies of NCWS patients. The researchers have just demonstrated a significant eosinophils infiltration of the duodenal and colon mucosa, and a significant infiltration of CD45+/CD3-CD14- cells in the rectal mucosa of NCWS patients upon wheat challenge, thus configuring a diffuse gastrointestinal "inflammatory/immunologic" pattern. As regard to rectal lymphocytes, analysis of cytokine production demonstrated dominant spontaneous interferon (IFN)-γ production by these cells, which were further identified as innate lymphoid cells belonging to the group 1 (ILC1) population, expressing T-bet and producing IFN-γ, compatible to an innate immunity involvement in NCWS pathogenesis. Therefore, the aims of the present study are: 1) to investigate the histological characteristics and differences in duodenal and rectal biopsies between NCWS and IBS patients, and 2) to search for "inflammatory/allergic" features (i.e. eosinophils and/or lymphocytes infiltration) useful for NCWS histological diagnosis.

ELIGIBILITY:
Inclusion Criteria:

To diagnose NCWS the recently proposed criteria will be adopted. All the patients will meet the following criteria:

* negative serum anti-transglutaminase (anti-tTG) and anti-endomysium (EmA) immunoglobulin (Ig)A and IgG antibodies
* absence of intestinal villous atrophy
* negative IgE-mediated immune-allergy tests to wheat (skin prick tests and/or serum specific IgE detection)
* resolution of the IBS symptoms on standard elimination diet, excluding wheat, cow's milk, egg, tomato, chocolate, and other self-reported food(s) causing symptoms
* symptom reappearance on double-blind placebo-controlled (DBPC) wheat challenge. As the investigators previously described in other studies, DBPC cow's milk protein challenge and other "open" food challenges will be performed too.

To diagnose IBS the standard Rome II (for retrospective patients) and Rome III (for prospective patients) Criteria will be adopted. None of these subjects improved on an elimination diet without wheat, cow's milk, egg, tomato, or chocolate.

Exclusion Criteria:

NCWS diagnosis will be excluded by:

* positive EmA in the culture medium of the duodenal biopsies, also in the case of normal villi/crypts ratio in the duodenal mucosa
* self-exclusion of wheat from the diet and refusal to reintroduce it before entering the study
* other previously diagnosed gastrointestinal disorders
* other previously diagnosed gynaecological disorders
* nervous system disease and/or major psychiatric disorder
* physical impairment limiting physical activity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include consecutive adult patients with IBS-like clinical presentation, according to Rome III criteria, and a definitive diagnosis of NCWS, referred at the Department of Internal Medicine at the University Hospital of Palermo, Italy, and at the Department of Internal Medicine of the Hospital of Sciacca, Agrigento, Italy, between July 2016 to February 2017, and sex- and age-matched subjects with IBS, enrolled at the same centers, as controls patients. All subjects will undergo upper gastrointestinal endoscopy and proctoscopy at the Gastroenterology Unit at the University Hospital of Palermo. Duodenal and rectal biopsies will be evaluated at 2 centers: the Pathology Unit at the University Hospital of Palermo, Italy, and the Institute of Pathology, Spedali Civili Brescia, Brescia, Italy.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Histological differences in duodenal biopsies between NCWS and IBS patients. | July 2016 to February 2017
  Histological characteristics and differences in duodenal biopsies between NCWS and IBS patients, with particular reference to lymphocytes, plasmacells, eosinophils and mast cells (i.e. number of cells for high power field).
Histological differences in rectal biopsies between NCWS and IBS patients. | July 2016 to February 2017
  Histological characteristics and differences in rectal biopsies between NCWS and IBS patients, with particular reference to lymphocytes, plasmacells, eosinophils and mast cells (i.e. number of cells for high power field).

SECONDARY OUTCOMES:
Identification of site (i.e. duodenal or rectal) with more inflammatory cells infiltration. | July 2016 to February 2017
  Evaluation of which examined site (i.e. duodenal or rectal) presents more lymphocytes and/or eosinophils infiltration (i.e. number of cells for high power field), for NCWS histological diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carroccio, PhD, Study Director — University of Palermo
Locations (2):
- Italy (2):
  - Department of Internal Medicine, Giovanni Paolo II Hospital of Sciacca, Sciacca, Agrigento
  - Department of Internal Medicine, University Hospital of Palermo, Palermo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carroccio A, Mansueto P, Iacono G, Soresi M, D'Alcamo A, Cavataio F, Brusca I, Florena AM, Ambrosiano G, Seidita A, Pirrone G, Rini GB. Non-celiac wheat sensitivity diagnosed by double-blind placebo-controlled challenge: exploring a new clinical entity. Am J Gastroenterol. 2012 Dec;107(12):1898-906; quiz 1907. doi: 10.1038/ajg.2012.236. Epub 2012 Jul 24. PMID 22825366
- [Result] Mansueto P, Seidita A, D'Alcamo A, Carroccio A. Non-celiac gluten sensitivity: literature review. J Am Coll Nutr. 2014;33(1):39-54. doi: 10.1080/07315724.2014.869996. PMID 24533607
- [Result] Carroccio A, Rini G, Mansueto P. Non-celiac wheat sensitivity is a more appropriate label than non-celiac gluten sensitivity. Gastroenterology. 2014 Jan;146(1):320-1. doi: 10.1053/j.gastro.2013.08.061. Epub 2013 Nov 22. No abstract available. PMID 24275240
- [Result] Carroccio A, D'Alcamo A, Mansueto P. Nonceliac wheat sensitivity in the context of multiple food hypersensitivity: new data from confocal endomicroscopy. Gastroenterology. 2015 Mar;148(3):666-7. doi: 10.1053/j.gastro.2014.11.047. Epub 2015 Jan 24. No abstract available. PMID 25625764
- [Result] Carroccio A, Soresi M, D'Alcamo A, Sciume C, Iacono G, Geraci G, Brusca I, Seidita A, Adragna F, Carta M, Mansueto P. Risk of low bone mineral density and low body mass index in patients with non-celiac wheat-sensitivity: a prospective observation study. BMC Med. 2014 Nov 28;12:230. doi: 10.1186/s12916-014-0230-2. PMID 25430806
- [Result] Mansueto P, Seidita A, D'Alcamo A, Carroccio A. Role of FODMAPs in Patients With Irritable Bowel Syndrome. Nutr Clin Pract. 2015 Oct;30(5):665-82. doi: 10.1177/0884533615569886. Epub 2015 Feb 18. PMID 25694210
- [Result] Di Liberto D, Mansueto P, D'Alcamo A, Lo Pizzo M, Lo Presti E, Geraci G, Fayer F, Guggino G, Iacono G, Dieli F, Carroccio A. Predominance of Type 1 Innate Lymphoid Cells in the Rectal Mucosa of Patients With Non-Celiac Wheat Sensitivity: Reversal After a Wheat-Free Diet. Clin Transl Gastroenterol. 2016 Jul 7;7(7):e178. doi: 10.1038/ctg.2016.35. PMID 27388423